CLINICAL TRIAL: NCT04162912
Title: Effects of a Motivational Interviewing Tailored Programme for Promoting Advance Care Planning Behaviours Among Patients With Palliative Care Needs: A Randomised Controlled Trial
Brief Title: Motivational Interviewing Tailored Programme for Promoting Advance Care Planning Behaviours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Health Bureau, Hong Kong (Other Government)
Collaborators: Haven of Hope Hospital (Other); United Christian Hospital (Other)
Responsible Party: Principal Investigator, Dr. Helen YL Chan, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14168417
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: End Stage Disease
Keywords: Advance Care Planning; Motivational Interviewing; Pallative Care

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group will receive a MotivationaI Interviewing tailored ACP programme.
  Interventions: Behavioral: Motivational Interviewing tailored Advance Care Planning
- Control group (No Intervention): The participants in the control group will receive usual care offered by the palliative care team under study and its affiliated day care centres, home care team and outpatient clinics.

INTERVENTIONS:
Behavioral: Motivational Interviewing tailored Advance Care Planning — The trained interventionist who is experienced in MI techniques will explore their illness experiences, emotions and beliefs about their health conditions and future care in an empathetic manner and explore their ambivalence for ACP behaviours.
  Arms: Experimental group

SUMMARY:
This proposed study is designed to test the effects of motivational interviewing (MI) in increasing the uptake of ACP behaviours among patients with palliative care needs. A randomised controlled trial with repeated blinded outcome assessment will be conducted to assess the effects of a MI-tailored ACP (MI-ACP) programme on palliative care patients recruited from the outpatient palliative care clinics and home palliative care services of two hospitals. A total of 204 patients will be recruited and randomly assigned to experimental and control groups. The patients in the experimental group will receive a MI-ACP programme facilitated by a trained nurse, whereas the patients in the control group will receive usual care. Primary outcome is the behavioural changes in ACP. Secondary outcomes are perceived stress, decisional conflict and quality of life. Study outcomes will be measured at baseline, 1 month and 3 months after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* newly referred to palliative care services
* with a palliative performance scale (PPS) score of 60 or above; and
* with full level of consciousness

Exclusion Criteria:

* uncommunicable because of sensory impairment or language barrier
* cognitively impaired
* are receiving active psychiatric treatment
* already had signed an advance directive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Advance Care Planning Behaviour | Baseline, 1 month and 3 months follow up
  Behaviour changes in ACP behaviours measured using a questionnaire. It included 4 items about different ACP behavior on a 5-point Likert scale. The higher score means the higher level of readiness for the behaviours.

SECONDARY OUTCOMES:
Decisional conflict | Baseline, 1 month and 3 months follow up
  Decisional conflict regarding end-of-life care is measured by the SURE test, a questionnaire with 4-item on knowledge and support for medical decision making. The higher score means the less decisional conflict.
Perceived stress | Baseline, 1 month and 3 months follow up
  Perceived stress is measured by a 10-item Perceived Stress Scale, a questionnaire, using a 5-point Likert scale. The higher score means the higher level of stress.
Quality of life | Baseline, 1 month and 3 months follow up
  Quality of life is measured by using a 23-item modified Quality of Life Concerns in the End of Life Questionnaire. The 23 items are rated on a 4-point Likert scale. The higher score means the better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Helen N Chan, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - United Christian Hospital, Kwun Tong
  - Haven of Hope Hospital, Tseung Kwan O

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan HY, Leung DY, Lam PT, Ko PP, Lam RW, Chan KS. Effect of motivational interviewing to promote advance care planning among palliative care patients in ambulatory care setting: a randomized controlled trial. BMC Palliat Care. 2025 Jan 31;24(1):31. doi: 10.1186/s12904-025-01667-9. PMID 39891169